CLINICAL TRIAL: NCT06533800
Title: VALUTAZIONE DEL MICROBIOTA E DEL RESISTOMA NEI DONATORI E NEI RICEVENTI DI FMT IN PAZIENTI CON INFEZIONE RICORRENTE DA CLOSTRIDIOIDES DIFFICILE
Brief Title: Evaluation of Gut Microbiota and Its Associated Resistome in FMT Donors and Recipients Due to Recurrent Clostridiodes Difficile Infection
Acronym: MICROFMT
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, De Maio Flavio, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6422
Record Dates: First submitted 2024-07-24; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: CDI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Caratterizzazione della composizione microbica intestinale nei donatori di FMT e nei pazienti affetti da rCDI al tempo basale e a seguito del trapianto di microbiota fecale. Negli stessi time point valutare il resistoma associato alla comunità microbica rilevata.

DETAILED DESCRIPTION:
Background Negli ultimi anni è diventata evidente l'importanza del microbioma intestinale nel mantenimento dell'omeostasi dell'individuo oltre che essere associato ad alcuni stati di malattia.

L'ospite e i microorganismi commensali costituiscono un sistema altamente integrato e dinamico che cambia in risposta a fattori ambientali (dieta, uso di farmaci o antibiotici, ambiente sociale) contribuendo al mantenimento dello stato di omeostasi o all'insorgenza di malattie [Reyman NatureCommunications 2022]. La comunità microbica intestinale è soggetta a cambiamenti fisiologici, nel corso della vita del singolo ospite, legati all'età [Aleman PlosPathogens 2019]. Negli ultimi anni, il trapianto di microbiota fecale (FMT) è diventato un approccio innovativo e promettente per trattare le infezioni ricorrenti da C. difficile (rCDI), con l'obiettivo di ripristinare una comunità microbica sana [Quaranta Journal of Applied Microbiology 2020]. Il maggiore utilizzo del FMT nella pratica clinica ha condotto a generare linee guida precise che descrivono le strutture e le procedure di laboratorio. Questo aspetto è particolarmente importante se si considera che la FMT è stata indicata per il trattamento di diverse patologie e non solo per la rCDI, per cui garantire la sicurezza del ricevente e monitorarne gli esiti sono alcuni degli obiettivi più importanti. In questo contesto, per ridurre al minimo il rischio di infezione o di trasmissione di altre malattie, i potenziali donatori sono sottoposti a uno screening rigoroso che comprende un'anamnesi approfondita, test sierologici e fecali per la ricerca di patogeni parassitari, virologici e batterici.

Razionale Mentre la valutazione del microbiota intestinale mediante analisi del 16s fornisce informazioni rapide sulla composizione microbica del donatore o sull'incidenza del ricevente, la caratterizzazione del resistoma potrebbe essere un altro parametro significativo da indagare.

L'intestino umano è una nicchia molto importante per i geni della resistenza antimicrobica (ARG) e il mobiloma, come insieme di elementi genetici che consentono il movimento di materiale genetico che alimenta il potenziale adattativo dei batteri, sebbene rimane ancora oscuro il suo impatto nella pratica clinica del FMT [Bargheet TheLancet 2023].

Nonostante il crescente numero di studi sulla FMT e sulle sue conseguenze nella risoluzione del rCDI, pochi o nessuno studio ha valutato i cambiamenti dinamici del microbiota intestinale e del resistoma, cercando contemporaneamente possibili fonti di ARG nei donatori e nei riceventi.

ELIGIBILITY:
Inclusion criteria

* patients with rCDI (> 18 years) to whom faecal microbiota transplantation is indicated, without other pathologies or prolonged hospitalization periods
* donors: healthy volunteers aged between 18 and 50 years
* Patients capable of expressing consent

Exclusion criteria

* antibiotic therapies in the last 30 days
* treatments with prebiotics - probiotics - postbiotics in the last 60 days
* colonization by MDR or XDR pathogens
* presence of pre-existing or ongoing intestinal pathologies (Inflammatory Intestinal Diseases, chronic hepatitis, celiac disease, neoplasms, previous large intestinal resections)
* ongoing diarrhea of any origin (defined as more than 6 watery stools per day and/or faecal volume greater than 250 ml in 24 hours)
* severe septic state in progress
* for donors: drug addiction, promiscuous sexual behaviour, use of drugs that can be excreted in the faeces with potential risk for recipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CDI patients - FMT donors
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of gut microbiota e associated resitome | 24 months
  Characterization of intestinal microbial composition in FMT donors and patients with rCDI at baseline time and following fecal microbiota transplantation. In the same time points evaluate the resistance associated with the microbial community detected.

IPD SHARING:
Plan to Share IPD: No